CLINICAL TRIAL: NCT04456634
Title: A Randomised, Single Blind, Placebo Controlled, Phase 1 Trial to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Activity of Ruxolitinib When Co-administered With Artemether-lumefantrine in Healthy Participants
Brief Title: Assess Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Profile of Ruxolitinib With Artemether-lumefantrine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Southern Star Research (Industry); Nucleus Network Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: MMV_Ruxolitinib_19_01
Record Dates: First submitted 2020-06-18; First posted 2020-07-02 (Actual); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Malaria
Keywords: Saftey; Tolerability
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination; ruxolitinib

STUDY DESIGN:
Intervention Model Description: 2 groups each to be enrolled sequentially. Group 1a will be a sentinel group of 2 participants, and Group 1b will be composed of 6 participants; to be administered either AL + Ruxolitinib or AL + placebo.
Who Masked: Participant
Masking Description: Randomised (single blinded; treatment allocation concealed to participants but not Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AL&RUX (Experimental): Oral administration of:
  • 20 mg/120 mg artemether-lumefantrine (AL) + 20 mg ruxolitinib phosphate (Rux)
  Interventions: Drug: 20 mg/120 mg artemether-lumefantrine (AL) + 20 mg ruxolitinib phosphate (Rux)
- AL& Placebo (Placebo Comparator): 20 mg/120 mg artemether-lumefantrine (AL) + Placebo
  Interventions: Other: 20 mg/120 mg artemether-lumefantrine (AL) + Placebo

INTERVENTIONS:
Drug: 20 mg/120 mg artemether-lumefantrine (AL) + 20 mg ruxolitinib phosphate (Rux) — Rux administered 2 hours after AL administration, twice daily (b.i.d) for 3 consecutive days (6 doses in total).
  Other Names: Sentinel Group 1 a and 1 b
  Arms: AL&RUX
Other: 20 mg/120 mg artemether-lumefantrine (AL) + Placebo — Placebo administered 2 hours after AL administration, twice daily (b.i.d) for 3 consecutive days (6 doses in total).
  Other Names: Sentinel Group 1 a and 1 b
  Arms: AL& Placebo

SUMMARY:
Phase 1, single -center study in 2 parts. The study designs for each part are well established for first-in-human studies and are appropriate to assess safety, tolerability and preliminary pharmacokinetics& pharmacodynamics.

DETAILED DESCRIPTION:
This is a randomised, single-blinded, placebo-controlled, single centre, phase 1 trial.

Eight healthy males or females, aged between 18-55 years old, who meet all of the inclusion criteria and none of the exclusion criteria, will be enrolled.

The study will be composed of 2 groups to be enrolled sequentially.

• Group 1a (sentinel group): two participants will be randomised single-blinded such that one participant will receive AL+Rux and the other participant will receive AL+placebo.

After review of the safety and tolerability data up to and including Day 8 from Group 1a by the Safety Review Committee (SRC), a decision to proceed with Group 1b will be made.

• Group 1b will be composed of 6 participants, to be randomised single-blinded such that five participants will receive AL+Rux, and one participant will receive AL+placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female (non-pregnant, non-lactating) aged 18 to 55 years inclusive.
2. Contactable and available for the duration of the trial and for up to two weeks following the EOS visit.
3. Total body weight greater than or equal to 50 kg, and a body mass index (BMI) within the range of 18 to 32 kg/m2 (inclusive) at Screening and Day -1. BMI is an estimate of body weight adjusted for height. It is calculated by dividing the weight in kilograms by the square of the height in metres.

   Health status
4. Certified as healthy by a comprehensive clinical assessment (detailed medical history, full physical examination and special investigations).
5. Vital signs measured after 5 min in the supine position:

   * Systolic blood pressure (SBP) - 90-140 mmHg,
   * Diastolic blood pressure (DBP) - 40-90 mmHg,
   * Heart rate (HR) 40-100 bpm.
6. ECG parameters for both males and females: QT ≤ 500 msec, QTcF ≤450 msec, QTcB ≤450 msec; PR interval ≤210 msec.
7. Heterosexual female participants of childbearing potential who have, or may have, male sexual partners during the course of the study should be using an insertable (implant or IUD), injectable, transdermal or combination oral contraceptive approved by the TGA combined with a barrier contraceptive from the time of informed consent until EOS. Abstinent female participants must agree to start a double method if they start a sexual relationship with a male during the trial. Female participants must not be planning in vitro fertilisation within the required contraception period.

   Women of non-childbearing potential who will not require contraception during the trial are defined as: surgically sterile (tubal ligation is not considered surgically sterile), post-menopausal (spontaneous amenorrhoea for ≥12 months, or spontaneous amenorrhoea for 6-12 months and follicle-stimulating hormone (FSH) ≥40 IU/mL; either should be together with the absence of oral contraceptive use for >12 months).

   Male participants who have, or may have female sexual partners during the course of the study must agree to use a double method of contraception including condom plus diaphragm, or condom plus stable insertable (implant or IUD), injectable, transdermal or combination oral contraceptive by the female partner, from the time of informed consent through to EOS. Abstinent male participants must agree to start a double method if they begin a sexual relationship with a female during the trial, and through to EOS. Male participants with female partners that are surgically sterile or post-menopausal, or male participants who have undergone sterilisation and have had testing to confirm the success of the sterilisation, may also be included and will not be required to use above described methods of contraception.

   Regulations
8. Completion of the written informed consent process prior to undertaking any trial-related procedure.
9. Must be willing and able to communicate and participate in the whole trial.
10. Agree to adhere to Lifestyle Considerations (see Section 4.3.3) throughout trial duration and be willing to consume 250 mL full-fat milk with each dose of AL.

Exclusion Criteria:

Medical history and clinical status

1. Known hypersensitivity to ruxolitinib, artesunate or any of its excipients, artemether, lumefantrine or other artemisinin derivatives, proguanil/atovaquone, primaquine, or 4-aminoquinolines.
2. Haematology, biochemistry or urinalysis results that are abnormal/outside of the laboratory normal reference ranges AND are either:

   * Considered clinically signficant by the Principal Investigator or delegate; OR
   * Considered not clinically significant by the Principal Investigator or delegate BUT ARE ALSO outside of Sponsor-approved clinically acceptable laboratory ranges in Appendix 1.

   NOTE: Participants are not excluded if abnormal/out of laboratory normal reference range results are considered not clinically significant by the Principal Investigator or delegate AND are within the ranges specified in Appendix 1.
3. Platelets < 200x109/L at Screening or prior to IMP administration is exclusionary. One re-test is permitted if original test result does not reflect the assumed medical status of the individual.
4. Participation in any other investigational product trial within 5 half-lives or 12 weeks preceding IMP administration, whichever is longer, or in the exclusion period of a previous trial according to applicable regulations.
5. Symptomatic postural hypotension at screening and pre-first dose of IMP on Day 1 (confirmed on two consecutive readings), irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 2-3 min when changing from supine to standing position.
6. History or presence of diagnosed (by an allergist/immunologist) or treated (by a physician) food or known drug allergies, or any history of anaphylaxis or other severe allergic reactions including face, mouth, or throat swelling or any difficulty breathing. Participants with seasonal allergies/hay fever or allergy to animals or house dust mite that are untreated and asymptomatic at the time of dosing can be enrolled in the trial.
7. History of convulsion (including drug or vaccine-induced episodes). A medical history of a single febrile convulsion during childhood is not an exclusion criterion.
8. Presence of current or suspected serious chronic diseases such as cardiac or autoimmune disease (HIV or other immuno-deficiencies), insulin-dependent and non-insulin-dependent diabetes, progressive neurological disease, severe malnutrition, acute or progressive hepatic disease, acute or progressive renal disease, porphyria, psoriasis, rheumatoid arthritis, asthma (excluding childhood asthma), epilepsy, or obsessive-compulsive disorder.
9. History of malignancy of any organ system (other than localised and considered cured basal cell carcinoma of the skin or in situ cervical cancer), treated or untreated, within five years of screening, regardless of whether there is no evidence of local recurrence or metastases.
10. Individuals with history of schizophrenia, bipolar disorder psychoses, disorders requiring lithium, attempted or planned suicide, or any other severe (disabling) chronic psychiatric diagnosis including generalised anxiety disorder.
11. Individuals who have been hospitalised within five years prior to enrolment for either a psychiatric illness or due to danger to self or others.
12. History of an episode of mild/moderate depression lasting more than 6 months that required pharmacological therapy and/or psychotherapy within the last 5 years; or any episode of major depression. The Beck Depression Inventory (BDI-II) will be used as a validated tool for the assessment of depression at screening. In addition to the conditions listed above, individuals with a score of 20 or more on the BDI-II and/or a response of 1, 2 or 3 for item 9 of this inventory (related to suicidal ideation) will not be eligible for participation. These individuals will be referred to a general practitioner or medical specialist as appropriate. Individuals with a BDI-II score of 17 to 19 may be enrolled at the discretion of an Investigator if they do not have a history of the psychiatric conditions mentioned in this criterion and their mental state is not considered to pose additional risk to the health of the individual or to the execution of the trial and interpretation of the data gathered.
13. History of recurrent headache (e.g. tension-type, cluster, or migraine) with a frequency of ≥2 episodes per month on average and severe enough to require medical therapy, during the 2 years preceding screening.
14. Acute illness within the 4 weeks prior to screening and prior to IMP administration.
15. Significant inter-current disease of any type, in particular liver, renal, cardiac, pulmonary, neurologic, rheumatologic, or autoimmune disease by history, physical examination, and/or laboratory studies including urinalysis.
16. Individual has a clinically significant disease or any condition or disease that might affect drug absorption, distribution or excretion (e.g. gastrectomy, cholecystectomy, diarrhoea) or known lactose/dairy intolerance.
17. Participation in any research trial involving blood sampling (more than 300 mL/unit of blood) within one month prior to IMP administration, or blood donation to Australian Red Cross Blood Service (Blood Service) or other blood bank during the 8 weeks prior to IMP administration.
18. Medical requirement for intravenous immunoglobulin or blood transfusions.
19. History or presence of alcohol abuse (alcohol consumption more than 40 g/4 units/4 standard drinks per day), or drug habituation, or any prior intravenous usage of an illicit substance.
20. Any individual who has ever smoked >1 pack of cigarettes per day for >10 years, or who currently (within 14 days prior to Screening or prior to IMP administration smokes >5 cigarettes/day.
21. Female who is breastfeeding.
22. Any vaccination within the last 28 days prior to screening or prior to IMP administration.
23. Prior to screening or IMP administration: any systemic or inhaled corticosteroids, anti-inflammatory drugs (excluding commonly used over-the-counter anti-inflammatory drugs such as ibuprofen, acetylsalicylic acid, diclofenac), immunomodulators or anticoagulants within the past three months. Any topical, nasal or ophthalmic corticosteroids within the past 2 weeks. Any individual currently receiving or having previously received immunosuppressive therapy (including systemic steroids, adrenocorticotrophic hormone or inhaled steroids) at a dose or duration potentially associated with hypothalamic-pituitary-adrenal axis suppression within the past year.
24. Use of antidepressant medication in the past 12 months prior to screening or prior to IMP administration.
25. Use of any other medication except contraceptives (including herbal, vitamin supplement, OTC or prescription) within 14 days or five half-lives (whichever is longest) prior to IMP administration. Participants areCONFIDENTIAL Page 7 of 78 requested to refrain from taking non-approved concomitant medications from recruitment until the conclusion of the trial.
26. Cardiac/QT risk:

    * Family history of sudden death or of congenital prolongation of the QTc interval or known congenital prolongation of the QTc interval or any clinical condition known to prolong the QTc interval.
    * History of symptomatic cardiac arrhythmias or with clinically relevant bradycardia.
    * Electrolyte disturbances, particularly hypokalaemia, hypocalcaemia, or hypomagnesaemia.
    * ECG abnormalities in the standard 12-lead ECG (at screening or prior to IMP administration) which in the opinion of an Investigator is clinically relevant or will interfere with the ECG analyses.

    General conditions
27. Any individual who, in the judgement of an Investigator, is likely to be non-compliant during the trial, or is unable to cooperate because of a language problem or poor mental development.
28. Any individual for whom study participation would pose an additional safety risk as assessed by the Principal Investigator.
29. Any individual who is an Investigator, research assistant, pharmacist, trial coordinator, or other staff thereof, directly involved in conducting the trial.
30. Any individual without good peripheral venous access. Biological status
31. Positive result on any of the following tests: hepatitis B surface antigen (HBs Ag), anti-hepatitis B core antibodies (anti-HBc Ab), anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti-HIV2 Ab).
32. Recent herpes zoster infection (within the previous 6 months) as determined by clinical history.
33. Positive result for M. tuberculosis infection by QuantiFERON-TB Gold assay.
34. Positive urine drug test for any drug listed in Section 7.4.5. Any individual testing positive for acetaminophen (paracetamol) at screening and/or pre-dose may still be eligible for trial participation at the discretion of the Principal Investigator or delegate.
35. Positive alcohol breath test.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Griffin, MD, Principal Investigator — Nucleus Network Corporate
Locations (1):
- Nucleus Network Brisbane, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chughlay MF, Barnes KI, El Gaaloul M, Abla N, Mohrle JJ, Griffin P, van Giersbergen P, Reuter SE, Schultz HB, Kress A, Tapley P, Webster RA, Wells T, McCarthy JS, Barber BE, Marquart L, Boyle MJ, Engwerda CR, Chalon S. Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Coadministered Ruxolitinib and Artemether-Lumefantrine in Healthy Adults. Antimicrob Agents Chemother. 2022 Jan 18;66(1):e0158421. doi: 10.1128/AAC.01584-21. Epub 2021 Oct 25. PMID 34694880

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 8 eligible participants were recruited at in the time period between 24 Aug 2020 and 19 Oct 2020 at Nucleus Network Brisbane clinic.
Pre-assignment Details: No wash out phase, no run-in phase. All eligible participants were dosed to the allocated doses on day 1. The study was composed of 2 groups to be enrolled sequentially.
Groups:
- AL&RUX: Oral administration of:
  • 20 mg/120 mg artemether-lumefantrine (AL) + 20 mg ruxolitinib phosphate (Rux)
  20 mg/120 mg artemether-lumefantrine (AL) + 20 mg ruxolitinib phosphate (Rux): Rux administered 2 hours after AL administration, twice daily (b.i.d) for 3 consecutive days (6 doses in total).
Period: Overall Study
Arm/Group | AL&RUX | AL& Placebo
Started | 6 | 2
Completed | 5 | 2
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AL&RUX | AL& Placebo | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 2 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.3 (11.8) | 30.0 (12.7) | 27.3 (27.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant With Treatment-Related Adverse Events as Assessed by CTCAE V4.03, All of Observed and Self-reported AEs Affected, by Treatment Regimen.
Description: Incidence, severity and relationship of observed and self-reported adverse events (AEs) were reported during the study up to 28 days after AL+Rux and AL+Placebo administration in all participants by treatment regimens.
Time Frame: up to 28 days after AL+Rux and AL+placebo administration
Population: All participants who received at least one dose of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | AL&RUX | AL& Placebo
Number analyzed (Participants) | 6 | 2
Participants | 6 | 2

2. Primary Outcome: Number of Participants With Changes of Systolic and Diastolic Blood Pressure
Description: Safety signals, trends or significant differences in blood pressure between treatment groups were were reported during the study up to 28 days after AL+Rux and AL+Placebo administration in all participants by treatment regimens.
Time Frame: up to 28 days after AL+Rux and AL+placebo administration
Population: All participants who received at least one dose of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | AL&RUX | AL& Placebo
Number analyzed (Participants) | 6 | 2
Participants | 2 | 0

3. Primary Outcome: Number of Participants With Changes in Heart Rate
Description: Safety signals, trends or significant differences in heart rate ( beats / min)between treatment groups were were reported during the study up to 28 days after AL+Rux and AL+Placebo administration in all participants by treatment regimens.
Time Frame: up to 28 days after AL+Rux and AL+placebo administration
Population: All participants who received at least one dose of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | AL&RUX | AL& Placebo
Number analyzed (Participants) | 6 | 2
Participants | 1 | 0

4. Primary Outcome: Number of Participants With ECG Changes
Description: Safety signals, trends or significant differences in QT, QTcB and QTcF, QRS between treatment groups were were reported during the study up to 28 days after AL+Rux and AL+Placebo administration in all participants by treatment regimens.
Time Frame: up to 28 days after AL+Rux and AL+placebo administration
Population: All participants who received at least one dose of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | AL&RUX | AL& Placebo
Number analyzed (Participants) | 6 | 2
Participants | 2 | 0

5. Secondary Outcome: AUECt of pSTAT3 Inhibition
Description: Area under the effect curve (AUECt) of pSTAT3 inhibition levels
Time Frame: up to 28 days after AL+Rux and AL+placebo administration
Population: All participants who received at least one dose of treatment
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Arm/Group | AL&RUX | AL& Placebo
Number analyzed (Participants) | 6 | 2
ng.hr/mL | 551 (86.9) | 186 (64.1)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from time of first dose of IMP until day 29 ( End of study visit) or early termination, approximately 29 days.
Arm/Group | AL&RUX | AL& Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 4/6 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AL&RUX (N=6) | AL& Placebo (N=2)
Muscular back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Vessel puncture site bruise (General disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
A PK drug-drug interaction between artemether and Rux cannot be excluded, and more data is needed to properly characterize such a potential interaction.

Investigation of possible PK drug-drug interactions were not within the scope of this study, due to small participant numbers, differing PK blood sampling schemes on Days 1 and 3, variability of artemether and lumefantrine PK parameters in the AL+Rux treatment group, and absence of a Rux-only treatment group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-07): https://cdn.clinicaltrials.gov/large-docs/34/NCT04456634/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/34/NCT04456634/SAP_001.pdf